CLINICAL TRIAL: NCT06614309
Title: Pilot Study to Investigate Possible Non-invasive Treatment for Long COVID (Post COVID-19 Condition) Brain Fog
Brief Title: Non-invasive Treatment for Long COVID (Post COVID-19 Condition) Brain Fog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney M. Wheatley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-006115
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Long COVID
Keywords: brain fog; brain blood flow; heart rate variability; fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Acute exposure: Placebo, Progressive Carbon Dioxide, Intermittent Hypoxia (Experimental): Study group will receive the three interventions in this order: Placebo, Progressive Carbon Dioxide, then Intermittent Hypoxia
  Interventions: Other: Acute Placebo Visit; Other: Acute Progressive Carbon Dioxide; Other: Acute Intermittent Hypoxia
- Acute exposure: Placebo, Intermittent Hypoxia, Progressive Carbon Dioxide (Experimental): Study group will receive the three interventions in this order: Placebo, Intermittent Hypoxia, Progressive Carbon Dioxide
  Interventions: Other: Acute Placebo Visit; Other: Acute Progressive Carbon Dioxide; Other: Acute Intermittent Hypoxia
- Acute exposure: Intermittent Hypoxia, Placebo, Progressive Carbon Dioxide (Experimental): Study group will receive the three interventions in this order: Intermittent Hypoxia, Placebo, Progressive Carbon Dioxide
  Interventions: Other: Acute Placebo Visit; Other: Acute Progressive Carbon Dioxide; Other: Acute Intermittent Hypoxia
- Acute exposure: Intermittent Hypoxia, Progressive Carbon Dioxide, Placebo (Experimental): Study group will receive the three interventions in this order: Intermittent Hypoxia, Progressive Carbon Dioxide, Placebo
  Interventions: Other: Acute Placebo Visit; Other: Acute Progressive Carbon Dioxide; Other: Acute Intermittent Hypoxia
- Acute exposure: Progressive Carbon Dioxide, Placebo, Intermittent Hypoxia (Experimental): Study group will receive the three interventions in this order: Progressive Carbon Dioxide, Placebo, Intermittent Hypoxia
  Interventions: Other: Acute Placebo Visit; Other: Acute Progressive Carbon Dioxide; Other: Acute Intermittent Hypoxia
- Acute exposure: Progressive Carbon Dioxide, Intermittent Hypoxia, Placebo (Experimental): Study group will receive the three interventions in this order: Progressive Carbon Dioxide, Intermittent Hypoxia, Placebo
  Interventions: Other: Acute Placebo Visit; Other: Acute Progressive Carbon Dioxide; Other: Acute Intermittent Hypoxia
- Placebo Group (Placebo Comparator): Study group will complete 6 simulated cycles of 5 minutes breathing 21% oxygen from a douglas bag and 5 minutes breathing room air (60 minutes) for every visit during the 14 days intervention period. Subjects will then return within 7 days of their final training visit to repeat baseline testing
  Interventions: Other: Training: Placebo Control
- Training Group (Experimental): Training Study group will be complete 6 cycles of either progressive CO2 ramp protocol or the intermittent hypoxia protocol for 60 minutes for every visit during the 14 days. Subjects will then return within 7 days of their final training visit to repeat baseline testing
  Interventions: Other: Training: Progressive Carbon Dioxide Ramping; Other: Training: Intermittent Hypoxic Exposure

INTERVENTIONS:
Other: Acute Placebo Visit — The placebo visit will include 6 simulated cycles of 5 minutes breathing 21% oxygen from a douglas bag and 5 minutes breathing room air.
  Arms: Acute exposure: Intermittent Hypoxia, Placebo, Progressive Carbon Dioxide; Acute exposure: Intermittent Hypoxia, Progressive Carbon Dioxide, Placebo; Acute exposure: Placebo, Intermittent Hypoxia, Progressive Carbon Dioxide; Acute exposure: Placebo, Progressive Carbon Dioxide, Intermittent Hypoxia; Acute exposure: Progressive Carbon Dioxide, Intermittent Hypoxia, Placebo; Acute exposure: Progressive Carbon Dioxide, Placebo, Intermittent Hypoxia
Other: Acute Progressive Carbon Dioxide — The progressive carbon dioxide visit will include a 60-minute progressive ramp which includes 6 cycles of progressive CO2 ramping starting at 0% and progressing up to 10% within 5 minutes immediately followed with 5 minutes of room air breathing in between cycles.
  Arms: Acute exposure: Intermittent Hypoxia, Placebo, Progressive Carbon Dioxide; Acute exposure: Intermittent Hypoxia, Progressive Carbon Dioxide, Placebo; Acute exposure: Placebo, Intermittent Hypoxia, Progressive Carbon Dioxide; Acute exposure: Placebo, Progressive Carbon Dioxide, Intermittent Hypoxia; Acute exposure: Progressive Carbon Dioxide, Intermittent Hypoxia, Placebo; Acute exposure: Progressive Carbon Dioxide, Placebo, Intermittent Hypoxia
Other: Acute Intermittent Hypoxia — The intermittent hypoxia exposure visit will include 6 cycles breathing 8-12% oxygen (O2) for 5 minutes with a target pulse oximeter saturation of 86-90%, followed by 5 minutes of breathing room air.
  Arms: Acute exposure: Intermittent Hypoxia, Placebo, Progressive Carbon Dioxide; Acute exposure: Intermittent Hypoxia, Progressive Carbon Dioxide, Placebo; Acute exposure: Placebo, Intermittent Hypoxia, Progressive Carbon Dioxide; Acute exposure: Placebo, Progressive Carbon Dioxide, Intermittent Hypoxia; Acute exposure: Progressive Carbon Dioxide, Intermittent Hypoxia, Placebo; Acute exposure: Progressive Carbon Dioxide, Placebo, Intermittent Hypoxia
Other: Training: Progressive Carbon Dioxide Ramping — Intervention will consist of 6 to 10 study visits (3-5 sessions/week) to be completed within 14 days. Subjects will will be given the progressive CO2 ramp protocol of 60-minute sessions, which will include 6 cycles of progressive CO2 ramping starting at 0% and progressing up to 10% within 5 minutes immediately followed with 5 minutes of room air breathing in between cycles, for every visit during the 14 days.
  Arms: Training Group
Other: Training: Intermittent Hypoxic Exposure — Intervention will consist of 6 to 10 study visits (3-5 sessions/week) to be completed within 14 days. Subjects will will be given the intermittent hypoxia exposure protocol of 60-minute sessions, which will include 6 cycles breathing 8-12% oxygen (O2) for 5 minutes with a target pulse oximeter saturation of 86-90%, followed by 5 minutes of breathing room air for every visit during the 14 days.
  Arms: Training Group
Other: Training: Placebo Control — Intervention will consist of 6 to 10 study visits (3-5 sessions/week) to be completed within 14 days. Subjects will complete 6 simulated cycles of 5 minutes breathing 21% oxygen from a douglas bag and 5 minutes breathing room air (60 minutes) for every visit during the 14 days.
  Arms: Placebo Group

SUMMARY:
This study aims to assess the effects of both acute and chronic exposures to hypoxia and hypercapnia in patients with Long COVID syndrome.

ELIGIBILITY:
Inclusion criteria:

* English speaking
* Diagnosis of Long COVID

Exclusion criteria:

* Any history of:

  * Coronary artery dissection or aortic dissection
  * Neurological disease (e.g. dementia, Alzheimer's disease, or other brain-related disease)
  * Cerebrovascular disease or stroke
  * Aneurysm
* If currently has:

  * Moderate-severe chronic obstructive pulmonary disease
  * Uncontrolled moderate-severe asthma
  * Moderate-severe bronchiectasis
  * Moderate-severe interstitial lung disease, requiring the use of supplemental oxygen
  * A necessity to use supplemental oxygen, for any reason
  * New or worsening symptoms (decompensation) of heart failure
  * Right heart disease due to chronic pulmonary disease/sleep apnea
  * Uncontrolled myocardial ischemia or angina
  * Uncontrolled heart arrhythmias
  * Heart or lung infection (e.g. myocarditis or pericarditis)
  * Left main coronary artery stenosis
  * Moderate-severe aortic stenosis
  * Pulmonary embolism, pulmonary infarction, or other blood clots
  * Severe respiratory disease
  * Chronic kidney disease
  * Chronic liver disease
* Females of childbearing potential will complete a urine pregnancy test at their baseline visit to rule out pregnancy
* BMI >40
* Study staff unable to obtain adequate signal for cerebral blood flow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral blood flow | Baseline, post-acute exposure and 14 days post training
  The intracranial middle cerebral arteries will be obtained (MCAv) will be imaged with a linear probe and duplex ultrasound system to simultaneously measure CBFv by pulse wave doppler (peak and mean flow)
Change in heart rate variability | Baseline, post-acute exposure and 14 days post training
  Short- term HRV analysis of a 3-lead ECG recording (5 minute recording) will evaluate both time-domain parameters (mean heart rate, standard deviation of normal-to-normal (NN) intervals (SDNN) and root mean square of successive differences between NN intervals rMSSD) and frequency-domain parameters (total power, high frequency (HF) and low frequency (LF) and LF/HF ratio).
Change in brain fog scale | Baseline, post-acute exposure and 14 days post training
  Questionnaire assessing of how much brain fog is affecting daily abilities

SECONDARY OUTCOMES:
Change in fatigue functional assessment of chronic illness therapy-fatigue scale | Baseline, post-acute exposure and 14 days post training
  Fatigue functional assessment of chronic illness therapy-fatigue scale (FACIT-Fatigue): assessment of how much fatigue is affecting daily abilities. Scores range from 0-52 for the FACIT with a higher score indicating higher levels of fatigue experienced.
Change in short form health survey (SF-36) | Baseline, post-acute exposure and 14 days post training
  The Short Form (SF-36) Health Survey is a 36-item, participant-reported survey that measures patient health and disability. Possible scores range from 0 to 100, with 0 indicating maximum disability, and 100 indicating no disability.
Change in Trail making test | Baseline, post-acute exposure and 14 days post training
  Trail making test: Consists of two parts. For part one, the subject will be presented with 25 numbered dots. The goal is to connect all 25 dots in numerical order quickly and accurately. The second part consists of 25 dots on the screen labelled with numbers and letters. The subject will then click the dots in sequential order by number followed by letter. For example, 1-A-2-B-3-C…, in the shortest amount of time possible while maintaining accuracy.
Change in rapid cognitive assessment tool (RCAT) score | Baseline, post-acute exposure and 14 days post training
  The premise is to click spawning targets quickly and accurately. The assessment lasts one minute during which the game will add or reduce intensity based on real time performance. It is used to interpret psychological and psychomotor functions including hand-eye coordination, speed, response time, spatial awareness, situational awareness, and decision-making. Test takes one minute and score is calculate based on number of correct clicks.
Change in Task switching test performance | Baseline, post-acute exposure and 14 days post training
  Task switching test will evaluate the individual's ability to switch between different tasks or operations. Participants are presented with a number between 1 and 9. The number will appear in one of two colors: purple or yellow. If the number is purple, the participant will answer with yes or no if the number is even. If yellow, the participants will answer with yes or no if the number is less than 5. Participants will see 40 numbers and their performance will be scored based on response time and accuracy.
Change in Rey Auditory Verbal Learning Test (AVLT) recall | Baseline, post-acute exposure and 14 days post training
  Rey Auditory Verbal Learning Test (AVLT) will assess short term auditory recall. Subjects are read a list of 15 words and asked to repeat as many words as possible that they can remember back to the test administrator. They repeat this 5 times, then read a new list of 15 words to repeat back one time before returning to recall the first list of words.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Wheatley-Guy, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No